CLINICAL TRIAL: NCT01777321
Title: Safety and Immunogenicity Study of GSK Biologicals' Herpes Zoster Subunit (HZ/su) Vaccine GSK1437173A When Administered Subcutaneously Versus Intramuscularly in Adults Aged 50 Years or Older
Brief Title: Safety and Immunogenicity Study of GSK Biologicals' Herpes Zoster Subunit (HZ/su) Vaccine GSK1437173A When Administered Subcutaneously Intramuscularly in Adults Aged ≥50 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 116760; 2012-005671-14 (EudraCT Number)
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-08

CONDITIONS: Herpes Zoster
Keywords: Herpes Zoster; Intramuscular; Subcutaneous; Safety; ≥50 years of age; Adults; Immunogenicity; Elderly
MeSH Terms: conditions — Herpes Zoster

ARMS (2):
- SC HZ/su Group (Experimental): Subjects will receive HZ/su vaccine administered SC on a 0,2-month schedule.
  Interventions: Biological: Herpes zoster vaccine GSK1437173A
- IM HZ/su Group (Active Comparator): Subjects will receive HZ/su vaccine administered IM on a 0,2-month schedule.
  Interventions: Biological: Herpes zoster vaccine GSK1437173A

INTERVENTIONS:
Biological: Herpes zoster vaccine GSK1437173A — HZ/su vaccine administered either into the subcutaneous tissue of the upper arm (deltoid region) of the non-dominant arm or intramuscularly in the deltoid region of non-dominant arm on a 0,2-month schedule.

SUMMARY:
The purpose of this study is to assess the immunogenicity, safety, and reactogenicity of GSK Biologicals' Herpes Zoster (HZ) vaccine (GSK 1437173A) when administered subcutaneously (SC) as compared to intramuscularly (IM) to people 50 years of age and older.

DETAILED DESCRIPTION:
There are 2 treatment groups in this study based upon the mode of vaccine administration.

The humoral immunogenicity (HI) will be measured in all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Subject, residing in Japan, is of Japanese ethnic origin, defined as having been born in Japan with four ethnic Japanese grandparents and able to speak Japanese.
* Subject has provided written informed consent.
* Subject, male or female, who is 50 YOA or older at the time of the first vaccination.
* Subject, if female, of non-childbearing potential may be enrolled in the study.
* Subject, if female, of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series (i.e., for 2 months after Month 2).
* Exclusion Criteria:
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Concurrently participating or planned participation in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Administration or planned administration of a live vaccine within 30 days prior to the first study vaccination through 30 days after the second study vaccination.
* Administration or planned administration of a non-replicating vaccine within 8 days prior to or within 14 days after either dose of study vaccine.
* Planned administration, during the study, of an HZ or varicella vaccine (including an investigational or non-registered vaccine) other than the study vaccine.
* Administration of immunoglobulins and/or any blood products within the three (3) months preceding the first dose of study vaccine or planned administration during the study period.
* Chronic administration (defined as >14 consecutive days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.

  * For corticosteroids, a prednisone dose of <20 mg/day, or equivalent, is allowed.
  * Inhaled, topical, and intra-articular corticosteroids are allowed.
* Administration or planned administration of long-acting immune-modifying drugs (e.g., infliximab) within six months prior to the first vaccine dose through the duration of the study period.
* History of HZ.
* Previous vaccination against HZ or varicella (registered or investigational product).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine or study material and equipment.
* Significant underlying illness that, in the opinion of the investigator, would be expected to prevent completion of the study.
* Any other condition that, in the opinion of the investigator, might interfere with the evaluations required by the study.
* Acute disease and/or fever at the time of vaccination:

  * Fever is defined as temperature ≥37.5°C (99.5°F) for oral, axillary, or tympanic route, or ≥38.0°C/100.4°F for rectal route. The preferred route for recording temperature in this study will be oral.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions (if of childbearing potential) through Month 4 (i.e., 2 months after the second dose of study vaccine).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06-17; Primary Completion 2013-10-10 (Actual); Study Completion 2014-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] de Oliveira Gomes J, Gagliardi AM, Andriolo BN, Torloni MR, Andriolo RB, Puga MEDS, Canteiro Cruz E. Vaccines for preventing herpes zoster in older adults. Cochrane Database Syst Rev. 2023 Oct 2;10(10):CD008858. doi: 10.1002/14651858.CD008858.pub5. PMID 37781954
- [Derived] Vink P, Shiramoto M, Ogawa M, Eda M, Douha M, Heineman T, Lal H. Safety and immunogenicity of a Herpes Zoster subunit vaccine in Japanese population aged >/=50 years when administered subcutaneously vs. intramuscularly. Hum Vaccin Immunother. 2017 Mar 4;13(3):574-578. doi: 10.1080/21645515.2016.1232787. Epub 2016 Dec 9. PMID 27936344
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 116760 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116760 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116760 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116760 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116760 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116760 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116760 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- SC GSK1437173A Group: Subjects received the GSK1437173A vaccine administered subcutaneously (SC) on a 0,2-month schedule.
- IM GSK1437173A Group: Subjects received the GSK1437173A vaccine administered intramuscularly (IM) on a 0,2-month schedule.
Period: Overall Study
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- SC GSK1437173A Group: Subjects received the GSK1437173A vaccine administered SC on a 0,2-month schedule.
- IM GSK1437173A Group: Subjects received the GSK1437173A vaccine administered IM on a 0,2-month schedule.
- Total: Total of all reporting groups
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.6 (7.59) | 62.2 (7.83) | 61.90 (7.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-Glycoprotein E (Anti-gE) Antibody Concentrations Higher Than or Equal to (≥)18 Milli-international Units Per Milliliter (mIU/mL)
Description: A seropositive subject was defined as a subject whose anti-gE Ab concentration was greater than or equal to the assay cut-off value, of 18 mIU/mL.
Time Frame: Before vaccination (PRE), two months after Dose 1 (M2) and one month after Dose 2 (M3)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects who had met all eligibility criteria and for whom data concerning immunogenicity outcome measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group
Number analyzed (Participants) | 29 | 29
Participants
  Anti-gE, PRE | 29 | 29
  Anti-gE, M2 | 29 | 29
  Anti-gE, M3 | 29 | 29

2. Primary Outcome: Anti-gE Antibody Concentrations
Description: Anti-gE antibody concentrations were expressed as geometric mean concentrations (GMCs) and measured in mIU/mL.
Time Frame: Before vaccination (PRE), two months after Dose 1 (M2) and one month after Dose 2 (M3)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects who had met all eligibility criteria and for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group
Number analyzed (Participants) | 29 | 29
mIU/mL
  Anti-gE, PRE | 1424.3 [1042.6 to 1945.6] | 1116.8 [774.5 to 1610.3]
  Anti-gE, M2 | 19902.5 [14846.9 to 26679.6] | 12842 [8558.4 to 19269.7]
  Anti-gE, M3 | 44126.1 [36326.1 to 53601] | 45521.5 [37549.5 to 55185.9]

3. Primary Outcome: Number of Subjects With Vaccine Response for Anti-gE Antibody Concentrations
Description: Vaccine response was defined as: For initially seronegative subjects, antibody concentration at post-vaccination ≥ 4 fold the cut-off for Anti-gE (4x18 mIU/mL); for initially seropositive subjects, antibody concentration at post-vaccination ≥ 4 fold the pre-vaccination antibody concentration.
Time Frame: At two months after Dose 1 (M2) and one month after Dose 2 (M3)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group
Number analyzed (Participants) | 29 | 29
Participants
  Anti-gE, M2 | 28 | 25
  Anti-gE, M3 | 29 | 29

4. Primary Outcome: Descriptive Statistics of Anti-gE Antibody Concentrations
Description: Anti-gE antibody concentrations were assessed by the Enzyme Lynked Immunosorbent Assay.
Time Frame: Before vaccination (PRE), at two months after dose 1 (M2) and one month after Dose 2 (M3)
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: mIU/mL
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group
Number analyzed (Participants) | 29 | 29
mIU/mL
  Anti-gE, PRE | 1404.1 (1398.82) | 946.3 (3231.78)
  Anti-gE, M2 | 19400.1 (24456.86) | 14330.1 (14548.75)
  Anti-gE, M3 | 44182 (27990.99) | 42444.8 (27555.21)

5. Primary Outcome: Number of Subjects With Solicited Local Symptoms
Description: The solicited local symptoms assessed were: Arm movement/range of motion of the vaccinated arm, Injection site pruritus, Pain, Redness, and Swelling. Any = occurrence of any local symptom regardless of their intensity grade. Grade 3 Pain = Significant pain at rest that prevented normal every day activities. Grade 3 Injection site pruritus = Significant pruritus that prevented normal every day activities. Grade 3 impairment of arm movement/range of motion = Significant impairment of arm movement/range of motion that prevented normal every day activities.
Time Frame: During the 7 day (Days 0-6) post vaccination, after each dose (D) and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one study vaccine administered and who had their symptom sheet filled-in.
Measure: Count of Participants; unit: Participants
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group
Number analyzed (Participants) | 30 | 30
Participants
  Any Arm movement impairment, D1 | 10 | 7
  Any Arm movement impairment, D2: number analyzed (Participants) | 30 | 29
  Any Arm movement impairment, D2 | 16 | 11
  Any Arm movement impairment, Across | 18 | 12
  Grade 3 Arm movement impairment, D1 | 1 | 0
  Grade 3 Arm movement impairment, D2: number analyzed (Participants) | 30 | 29
  Grade 3 Arm movement impairment, D2 | 0 | 0
  Grade 3 Arm movement impairment, Across | 1 | 0
  Any Injection site pruritus, D1 | 19 | 6
  Any Injection site pruritus, D2: number analyzed (Participants) | 30 | 29
  Any Injection site pruritus, D2 | 15 | 8
  Any Injection site pruritus, Across | 21 | 10
  Grade 3 Injection site pruritus, D1 | 0 | 0
  Grade 3 Injection site pruritus, D2: number analyzed (Participants) | 30 | 29
  Grade 3 Injection site pruritus, D2 | 0 | 0
  Grade 3 Injection site pruritus, Across | 0 | 0
  Any Pain, D1 | 28 | 26
  Any Pain, D2: number analyzed (Participants) | 30 | 29
  Any Pain, D2 | 25 | 21
  Any Pain, Across | 28 | 27
  Grade 3 Pain, D1 | 2 | 0
  Grade 3 Pain, D2: number analyzed (Participants) | 30 | 29
  Grade 3 Pain, D2 | 1 | 0
  Grade 3 Pain, Across | 2 | 0
  Any Redness, D1 | 23 | 11
  Any Redness, D2: number analyzed (Participants) | 30 | 29
  Any Redness, D2 | 23 | 12
  Any Redness, Across | 26 | 15
  Grade 3 Redness, D1 | 12 | 1
  Grade 3 Redness, D2: number analyzed (Participants) | 30 | 29
  Grade 3 Redness, D2 | 12 | 1
  Grade 3 Redness, Across | 17 | 2
  Any Swelling, D1 | 22 | 7
  Any Swelling, D2: number analyzed (Participants) | 30 | 29
  Any Swelling, D2 | 20 | 11
  Any Swelling, Across | 24 | 12
  Grade 3 Swelling, D1 | 8 | 1
  Grade 3 Swelling, D2: number analyzed (Participants) | 30 | 29
  Grade 3 Swelling, D2 | 6 | 1
  Grade 3 Swelling, Across | 10 | 2

6. Primary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were: Fatigue, Fever, Gastrointestinal (nausea, vomiting, diarrhea and/or abdominal pain), Headache, Myalgia, and Shivering. Fever = axillary temperature ≥37.5°C. Any = occurrence of any general symptoms regardless of their intensity grade or relationship to vaccination. Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 Fever = axillary temperature higher than (>) 39.0°C. Related = general symptom assessed by the investigator as causally related to vaccination.
Time Frame: During the 7 day (Days 0-6) post vaccination, after each dose (D) and across doses
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group
Number analyzed (Participants) | 30 | 30
Participants
  Any Fatigue, D1 | 14 | 12
  Any Fatigue, D2: number analyzed (Participants) | 30 | 29
  Any Fatigue, D2 | 16 | 9
  Any Fatigue, Across | 21 | 16
  Grade 3 Fatigue, D1 | 0 | 0
  Grade 3 Fatigue, D2: number analyzed (Participants) | 30 | 29
  Grade 3 Fatigue, D2 | 0 | 1
  Grade 3 Fatigue, Across | 0 | 1
  Related Fatigue, D1 | 14 | 12
  Related Fatigue, D2: number analyzed (Participants) | 30 | 29
  Related Fatigue, D2 | 16 | 9
  Related Fatigue, Across | 21 | 16
  Any Fever/Axillary, D1 | 3 | 2
  Any Fever/Axillary, D2: number analyzed (Participants) | 30 | 29
  Any Fever/Axillary, D2 | 5 | 6
  Any Fever/Axillary, Across | 6 | 7
  Grade 3 Fever/Axillary, D1 | 0 | 0
  Grade 3 Fever/Axillary, D2: number analyzed (Participants) | 30 | 29
  Grade 3 Fever/Axillary, D2 | 0 | 0
  Grade 3 Fever/Axillary, Across | 0 | 0
  Related Fever/Axillary, D1 | 3 | 2
  Related Fever/Axillary, D2: number analyzed (Participants) | 30 | 29
  Related Fever/Axillary, D2 | 5 | 6
  Related Fever/Axillary, Across | 6 | 7
  Any Gastrointestinal symptoms, D1 | 2 | 4
  Any Gastrointestinal symptoms, D2: number analyzed (Participants) | 30 | 29
  Any Gastrointestinal symptoms, D2 | 5 | 3
  Any Gastrointestinal symptoms, Across | 7 | 5
  Grade 3 Gastrointestinal symptoms, D1 | 0 | 0
  Grade 3 Gastrointestinal symptoms, D2: number analyzed (Participants) | 30 | 29
  Grade 3 Gastrointestinal symptoms, D2 | 0 | 1
  Grade 3 Gastrointestinal symptoms,Across | 0 | 1
  Related Gastrointestinal symptoms, D1 | 2 | 4
  Related Gastrointestinal symptoms, D2: number analyzed (Participants) | 30 | 29
  Related Gastrointestinal symptoms, D2 | 5 | 3
  Related Gastrointestinal symptoms,Across | 7 | 5
  Any Headache, D1 | 11 | 8
  Any Headache, D2: number analyzed (Participants) | 30 | 29
  Any Headache, D2 | 11 | 10
  Any Headache, Across | 17 | 13
  Grade 3 Headache, D1 | 0 | 0
  Grade 3 Headache, D2: number analyzed (Participants) | 30 | 29
  Grade 3 Headache, D2 | 0 | 2
  Grade 3 Headache, Across | 0 | 2
  Related Headache, D1 | 11 | 8
  Related Headache, D2: number analyzed (Participants) | 30 | 29
  Related Headache, D2 | 11 | 10
  Related Headache, Across | 17 | 13
  Any Myalgia, D1 | 2 | 1
  Any Myalgia, D2: number analyzed (Participants) | 30 | 29
  Any Myalgia, D2 | 5 | 3
  Any Myalgia, Across | 7 | 4
  Grade 3 Myalgia, D1 | 1 | 0
  Grade 3 Myalgia, D2: number analyzed (Participants) | 30 | 29
  Grade 3 Myalgia, D2 | 0 | 1
  Grade 3 Myalgia, Across | 1 | 1
  Related Myalgia, D1 | 2 | 1
  Related Myalgia, D2: number analyzed (Participants) | 30 | 29
  Related Myalgia, D2 | 5 | 3
  Related Myalgia, Across | 7 | 4
  Any Shivering, D1 | 3 | 3
  Any Shivering, D2: number analyzed (Participants) | 30 | 29
  Any Shivering, D2 | 6 | 6
  Any Shivering, Across | 8 | 7
  Grade 3 Shivering, D1 | 0 | 1
  Grade 3 Shivering, D2: number analyzed (Participants) | 30 | 29
  Grade 3 Shivering, D2 | 0 | 0
  Grade 3 Shivering, Across | 0 | 1
  Related Shivering, D1 | 3 | 3
  Related Shivering, D2: number analyzed (Participants) | 30 | 29
  Related Shivering, D2 | 6 | 6
  Related Shivering, Across | 8 | 7

7. Primary Outcome: Mean Number of Days With Local Symptoms
Description: Days with solicited local symptoms were tabulated for the total vaccinated cohort.
Time Frame: During the 7 day (Days 0-6) post vaccination, after each dose (D)
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one study vaccine administered.
Measure: Mean (Inter-Quartile Range); unit: Days
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group
Number analyzed (Participants) | 30 | 30
Days
  Days with arm movement, D1 | 3.9 [2 to 7] | 3 [2 to 3]
  Days with pain, D1 | 3.3 [2 to 4] | 2.7 [2 to 3]
  Days with injection site pruritus, D1 | 5.2 [2 to 7] | 2.2 [1 to 3]
  Days with redness, D1 | 6.5 [4 to 8] | 2.6 [2 to 3]
  Days with swelling, D1 | 5 [3 to 6] | 3 [2 to 3]
  Days with arm movement, D2 | 2.9 [2 to 3] | 2.2 [2 to 3]
  Days with pain, D2 | 3.4 [2 to 4] | 2.3 [1 to 3]
  Days with injection site pruritus, D2 | 4.9 [3 to 5] | 1.9 [1.5 to 2]
  Days with redness, D2 | 5.9 [3 to 6] | 3.7 [3 to 4]
  Days with swelling, D2 | 4.3 [3 to 6] | 2.8 [2 to 4]

8. Primary Outcome: Mean Number of Days With General Symptoms
Description: Days with solicited general symptoms were tabulated for the total vaccinated cohort.
Time Frame: During the 7 day (Days 0-6) post vaccination, after each dose (D)
Population: as for outcome 7
Measure: Mean (Inter-Quartile Range); unit: Days
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group
Number analyzed (Participants) | 30 | 30
Days
  Days with fatigue, D1 | 2.3 [1 to 3] | 2 [1 to 2]
  Days with fever, D1 | 1.3 [1 to 2] | 1 [1 to 1]
  Days with gastrointestinal symptoms, D1 | 2 [1 to 3] | 2 [2 to 2]
  Days with headache, D1 | 1.8 [1 to 2] | 1.4 [1 to 2]
  Days with myalgia, D1 | 6.5 [3 to 10] | 2 [2 to 2]
  Days with Shivering, D1 | 1.3 [1 to 2] | 1.3 [1 to 2]
  Days with fatigue, D2 | 2 [1 to 2] | 1.3 [1 to 2]
  Days with fever, D2 | 1 [1 to 1] | 1 [1 to 1]
  Days with gastrointestinal symptoms, D2 | 3.6 [2 to 5] | 1.3 [1 to 2]
  Days with headache, D2 | 2 [1 to 2] | 1.3 [1 to 2]
  Days with myalgia, D2 | 2 [1 to 2] | 1.3 [1 to 2]
  Days with Shivering, D2 | 2.2 [1 to 2.2] | 1 [1 to 1]

9. Primary Outcome: Number of Subjects With Potential Immune-Mediated Disorders (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) were a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From Month 0 to Month 3
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

10. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within 30 days (Days 0-29) post vaccination period
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group
Number analyzed (Participants) | 30 | 30
Participants
  Any AEs | 9 | 6
  Grade 3 AEs | 1 | 0
  Related AEs | 1 | 1

11. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Month 0 to Month 3
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group
Number analyzed (Participants) | 30 | 30
Participants | 1 | 0

12. Secondary Outcome: Number of Subjects With Anti-gE Antibody Concentrations ≥ 97 mIU/mL
Description: A seropositive subject was defined as a subject whose anti-gE Ab concentration was greater than or equal to the assay cut-off value of 97 mIU/mL.
Time Frame: At Month 14
Population: The analysis was performed on the ATP cohort for persistence, which included all evaluable subjects for whom data concerning immunogenicity persistence outcome variables were available.
Measure: Count of Participants; unit: Participants
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group
Number analyzed (Participants) | 30 | 28
Participants | 30 | 28

13. Secondary Outcome: Anti-gE Antibody Concentrations
Description: Anti-gE antibody concentrations were expressed as geometric mean concnetrations (GMCs) and measured in mIU/mL.
Time Frame: At Month 14
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group
Number analyzed (Participants) | 30 | 30
mIU/mL | 15250.9 [12464 to 18660.9] | 13870.2 [10184.2 to 18890.3]

14. Secondary Outcome: Number of Subjects With Vaccine Response for Anti-gE Antibody Concentrations
Description: Vaccine response was defined as: For initially seronegative subjects, antibody concentration at post-vaccination ≥ 4 fold the cut-off for Anti-gE (4x97 mIU/mL); for initially seropositive subjects, antibody concentration at post-vaccination ≥ 4 fold the pre-vaccination antibody concentration.
Time Frame: Twelve Months after Dose 2 (M14)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group
Number analyzed (Participants) | 30 | 28
Participants | 25 | 25

15. Secondary Outcome: Number of Subjects With pIMDs
Description: as for outcome 9
Time Frame: Up to Month 14 post vaccination period
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

16. Secondary Outcome: Number of Subjects With SAEs
Description: as for outcome 11
Time Frame: Up to Month 14 post vaccination period
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group
Number analyzed (Participants) | 30 | 30
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 7-day post-vaccination period; Unsolicited AEs: during the 30-day post-vaccination period; SAEs: up to Month 14 post vaccination.
Description: No unsolicited AEs with a frequency over 5% were reported.
Arm/Group | SC GSK1437173A Group | IM GSK1437173A Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 2/30 | 1/30
Other Adverse Events (participants affected / at risk) | 30/30 | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SC GSK1437173A Group (N=30) | IM GSK1437173A Group (N=30)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mallet finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SC GSK1437173A Group (N=30) | IM GSK1437173A Group (N=30)
Arm movement (General disorders) | 18 (18) | 12 (12)
Injection site pruritus (General disorders) | 21 (21) | 10 (10)
Pain (General disorders) | 28 (28) | 27 (27)
Redness (General disorders) | 26 (26) | 15 (15)
Swelling (General disorders) | 24 (24) | 12 (12)
Fatigue (General disorders) | 21 (21) | 16 (16)
Fever/(Axillary) (General disorders) | 6 (6) | 7 (7)
Gastrointestinal symptoms (General disorders) | 7 (7) | 5 (5)
Headache (General disorders) | 17 (17) | 13 (13)
Myalgia (muscle aches) (General disorders) | 7 (7) | 4 (4)
Shivering (General disorders) | 8 (8) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.